CLINICAL TRIAL: NCT00453869
Title: Screening of Fibrosing and/or Viral Chronic Hepatopathies in Jail
Acronym: SNIFF11
Status: Terminated | Type: Observational
Why Stopped: Few prevalence of liver fibrosis in subjects
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC 2006-05; DGS 2006-0142 ; CPP 2006/27bis
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Liver Fibrosis
Keywords: Liver fibrosis; Hepatitis B virus and C virus; FibroMeter; FibroScan®
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: liver fibrosis evaluation — Evaluation of liver fibrosis with blood test

SUMMARY:
The prevalence of chronic hepatopathies is high in jail. However, the medical care of these hepatopathies is few developed. This study is an observational, an epidemiologic (screening and prevalence of fibrosing hepatopathies) and an evaluating study for a better taking care of these hepatopathies in jail. The aims of the study will be to evaluate the diagnostic performance of the FibroMeter score in the screening of the hepatic fibrosis in persons with multiple risk factors for liver fibrosis (alcoholism, intravenous drug users, tattoo, and virological status) with FibroScan® as gold standard; to evaluate the feasibility of these different screening tools for chronic hepatopathies in jail and to evaluate the prevalence of the fibrosing hepatopathies with clinically significant fibrosis and theirs risk factors, alcohol and hepatitis B and hepatitis C viruses in population from Angers jail.

DETAILED DESCRIPTION:
Primary outcome: Screening of clinically significant fibrosis with FibroMeter blood score. Screening for hepatitis B and hepatitis C viruses.

Secondary outcome: Clinically significant fibrosis confirmed with FibroScan®.

The means for this study are a clinical questionnaire, a virological screening, a blood score for liver fibrosis: FibroMeter according to cause of the fibrosis and FibroScan® is referent and independent examination.

The expected results from this study are the knowledge of the prevalence of hepatopathies with hepatic fibrosis will be able to justify, possibly, a screening politic of them. This study will permit to evaluate the feasibility of noninvasive screening of the liver fibrosis in the goal to suppress the liver biopsy in a population having numerous drawbacks.

ELIGIBILITY:
Inclusion Criteria:

* Person over 18,
* All new inmates, for less than one month, in Angers jail,
* To have a written informed consent.

Exclusion Criteria:

* No consent obtained from person,
* Detention inferior to one month,
* Person under 18.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects in jail who have a medical evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Liver fibrosis evaluation | D0
  Evaluation of liver fibrosis with blood tests

CONTACTS AND LOCATIONS:
Overall Officials: Paul CALES, MD, PhD, Principal Investigator — UH Angers
Locations (1):
- University Hospital Angers, Angers, France